CLINICAL TRIAL: NCT02893267
Title: Multimodal Treatment for Hemiplegic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Case Western Reserve University (Other); Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Richard Wilson, MD, Assistant Professor, Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB16-00172; R01HD084564 (NIH)
Record Dates: First submitted 2016-08-31; First posted 2016-09-08 (Estimated); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Shoulder Pain
Keywords: Stroke; Shoulder Pain; Electrical stimulation; Neuromuscular stimulation; Intramuscular stimulation; Physical Therapy
MeSH Terms: conditions — Stroke; Shoulder Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- PNS + PT (Experimental): The PNS+PT Group will receive peripheral nerve stimulation treatment (which will produce muscle contraction) for three weeks (6 hours daily) with an Intramuscular Electrical Stimulator following a one week electrode stabilization period, and also receive eight 60-minute sessions of outpatient physical therapy focused on shoulder pain over the same four week period.
  Interventions: Device: Peripheral Nerve Stimulation; Other: Physical Therapy
- PNS + sham-PT (Active Comparator): The PNS + sham-PT Group will receive peripheral nerve stimulation treatment (which will produce muscle contraction) for three weeks (6 hours daily) with an Intramuscular Electrical Stimulator following a one week electrode stabilization period, and also receive eight 60-minute sessions of sham outpatient physical therapy not focused on shoulder pain over the same four week period.
  Interventions: Device: Peripheral Nerve Stimulation; Other: Sham-PT
- sham-PNS + PT (Active Comparator): The sham-PNS + PT Group will receive sham peripheral nerve stimulation treatment (which will not produce muscle contraction) for three weeks (6 hours daily) with an Intramuscular Electrical Stimulator following a one week electrode stabilization period, and also receive eight 60-minute sessions of outpatient physical therapy focused on shoulder pain over the same four week period.
  Interventions: Other: Physical Therapy; Device: Sham-PNS

INTERVENTIONS:
Device: Peripheral Nerve Stimulation — The stimulation system includes an external stimulator, percutaneous lead and pad. The stimulator snaps onto the pad. The pad has an embedded power source but also serves as the anode. The 1-channel stimulator outputs a biphasic current waveform with current pulse parameter ranges suitable for PNS. The percutaneous lead is inserted using an introducer (like a hypodermic needle) which is withdrawn and the lead is retained in the muscle by a barb at its tip. After a 1-week stabilization period, stimulation is initiated (6 hrs/day). The duty cycle and daily dose remain constant, but stimulus parameters may be adjusted by the research staff as deemed appropriate. The treatment period is 3 weeks after which the lead will be removed. Total time of electrode implantation is no more than 29 days.
  Other Names: Intramuscular Peripheral Nerve Stimulation; Intramuscular Electrical Nerve Stimulation; Smartpatch System
  Arms: PNS + PT; PNS + sham-PT
Other: Physical Therapy — Participants will receive 8 60-minute sessions of outpatient therapy over a 4 week period concurrent with PNS or sham-PNS treatment. Therapy may include: Proper Positioning and Handling, Therapeutic positioning and Strengthening Exercises, Mirror Therapy, Task-specific Therapy, Home Exercise Program, and a Mental Practice program.
  Arms: PNS + PT; sham-PNS + PT
Other: Sham-PT — Participants randomized to sham-PT will receive 8 60-minute sessions with therapists with the goal of controlling for the effect of regular contact with a therapist and study staff in a therapeutic environment. Participants will undergo a hands-on evaluation and re-evaluation before and after treatment. Therapists will provide sham ultrasound therapy and light application of inert gel to the shoulder for 10 minutes, Pre-Gait Training or Gait training, Exercise therapy, and relaxation therapy.
  Arms: PNS + sham-PT
Device: Sham-PNS — The stimulation system includes an external stimulator, percutaneous lead and pad. The stimulator snaps onto the pad. The pad has an embedded power source.The stimulator will appear to function as normal though will not deliver electrical current to the electrode. The subjects will be prescribed 6 hours of sham-stimulation per day for 3 weeks.
  Arms: sham-PNS + PT

SUMMARY:
Hemiplegic shoulder pain (HSP) affects up to 60% of moderate to severely impaired stroke survivors. HSP is associated with poor rehabilitation outcomes, including interference with activities of daily living (ADLs) and poor quality of life (QoL). While many treatments for HSP have been proposed, most do not result in long-term relief of pain.

The investigators developed the use of intramuscular peripheral nerve stimulation (PNS) for the treatment of HSP, which involves the temporary placement of a percutaneous intramuscular electrode to stimulate the axillary nerve motor points to the deltoid muscle. A systematic review of randomized controlled trials (RCT) concluded that intramuscular PNS was the only treatment to provide long-term relief of pain for those with HSP. However, physical therapy (PT), which focuses on correcting biomechanics, is the most commonly prescribed treatment for HSP and is recommended by multiple practice guidelines. Prior to acceptance by the clinical community, the superiority of PNS to a course of PT must be demonstrated. The investigators completed a pilot RCT comparing PNS to PT and 67% vs. 25% of participants experienced successful pain relief (i.e., ≥ 2-pt or 30% reduction) from PNS and PT, respectively. Thus, the primary objective of this 2-site RCT is to confirm the findings of this preliminary pilot RCT. Combining PNS and PT, which may be how PNS is actually implemented in clinical practice, may have a synergistic therapeutic effect. Thus, the second objective of this RCT is to determine if multimodal treatment of HSP with PNS + PT is more efficacious for pain relief than PNS alone or PT alone. Mechanisms also will be explored.

DETAILED DESCRIPTION:
Study Summary: This is a multi-site, placebo controlled, double-blinded RCT to confirm the superiority of PNS over PT in reducing HSP, and to determine if multimodal treatment of HSP with PNS + PT is more efficacious than PNS or PT alone. The standard of care for treating shoulder pain is to try several options, most commonly including medications, injections and therapy. Candidates considering this study likely have tried some treatments but without lasting success. Ninety-six participants will be randomized to receive PNS + PT, PNS + sham-PT, or sham-PNS + PT. The PNS + PT group will receive active PNS therapy for 6 hours per day for 3 weeks along with 8 sessions of PT to improve biomechanics of the affected shoulder. The PNS+ sham-PT group will receive active PNS therapy and sham-PT, consisting of placebo ultrasound, application of inert gel, lower limb strengthening, and walking exercises. The sham-PNS + PT group will receive a percutaneous lead in a similar manner as the active therapy groups, but with sham-stimulation, along with 8 sessions of PT. Measures of pain, pain interference with ADLs, QoL, shoulder biomechanics (shoulder abduction torque, shoulder kinematics, and Fugl-Meyer score), and measures of central sensitization (pain thresholds, secondary hyperalgesia, and temporal summation) will be assessed at baseline and at weeks 4 (end of treatment), 8, 12, 16, 20, 24, and 28.

ELIGIBILITY:
Inclusion Criteria:

* shoulder pain localized to the glenohumeral joint, subacromial area or deltoid insertion associated with: a) rest; b) passive abduction or external rotation range of motion (ROM); c) active abduction ROM; or, d) manual palpation;
* shoulder pain onset or worsening after the most recent stroke;
* weakness of shoulder abductors (≤4/5 on Medical Research Council (MRC) scale if isolated movement is present);
* ≥ 21-yrs old; < 90-yrs old;
* time of stroke ≥ 3-mo;
* duration of HSP ≥3-mo;
* HSP with moderate to severe pain (BPI SF-3 ≥ 4);
* cognitive and communication ability to fulfill study requirements (cognitive ability based upon a score of ≥24 on the Mini Mental Status Exam (MMSE));
* availability of reliable adult who can assist with study procedures if necessary;
* willing and able to report shoulder pain and other conditions and complete study visits throughout the 4 month study period.

Exclusion Criteria:

* joint or overlying skin infection or history of recurrent skin infections;
* insensate skin;
* need to take > 1 opioid and > 1 nonopioid analgesic medication for HSP;
* regular intake of pain medications for another chronic pain;
* botox injection or subacromial steroid injections to the shoulder within the past 12 weeks;
* receiving occupational therapy (OT) or PT for HSP;
* bleeding disorder or international normalized ratio (INR) > 3.0;
* sensitivity to skin surface electrodes and/or medical-grade adhesives, gels, tapes;
* medical instability;
* pregnancy;
* uncontrolled seizures (>1/mo for 6-mo);
* history of cardiac arrhythmia with hemodynamic instability;
* history of lidocaine allergy;
* history of Parkinson's disease, spinal cord injury (SCI), traumatic brain injury (TBI), multiple sclerosis (MS), or ipsilateral upper extremity (UE) lower motor neuron lesion;
* history of complex regional pain syndrome, myofacial pain syndrome, other pain conditions (investigator discretion);
* cardiac pacemaker or other implanted electronic device;
* history of valvular heart disease (artificial valves, requiring antibiotics for procedures, etc.);
* severely impaired communication.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-01; Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Wilson, MD, Principal Investigator — MetroHealth Medical Center
Locations (3):
- United States (3):
  - Shirley Ryan Abilitylab, Chicago, Illinois
  - Carolinas Rehabilitation, Charlotte, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson RD, Gunzler DD, Bennett ME, Chae J. Peripheral nerve stimulation compared with usual care for pain relief of hemiplegic shoulder pain: a randomized controlled trial. Am J Phys Med Rehabil. 2014 Jan;93(1):17-28. doi: 10.1097/PHM.0000000000000011. PMID 24355994
- [Background] Chae J, Ng A, Yu DT, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Fang ZP. Intramuscular electrical stimulation for shoulder pain in hemiplegia: does time from stroke onset predict treatment success? Neurorehabil Neural Repair. 2007 Nov-Dec;21(6):561-7. doi: 10.1177/1545968306298412. Epub 2007 Mar 16. PMID 17369520
- [Background] Chae J, Wilson RD, Bennett ME, Lechman TE, Stager KW. Single-lead percutaneous peripheral nerve stimulation for the treatment of hemiplegic shoulder pain: a case series. Pain Pract. 2013 Jan;13(1):59-67. doi: 10.1111/j.1533-2500.2012.00541.x. Epub 2012 Mar 26. PMID 22448759
- [Background] Chae J, Yu D, Walker M. Percutaneous, intramuscular neuromuscular electrical stimulation for the treatment of shoulder subluxation and pain in chronic hemiplegia: a case report. Am J Phys Med Rehabil. 2001 Apr;80(4):296-301. doi: 10.1097/00002060-200104000-00014. PMID 11277137
- [Background] Chae J, Yu DT, Walker ME, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Frost FS, Grill JH, Fang ZP. Intramuscular electrical stimulation for hemiplegic shoulder pain: a 12-month follow-up of a multiple-center, randomized clinical trial. Am J Phys Med Rehabil. 2005 Nov;84(11):832-42. doi: 10.1097/01.phm.0000184154.01880.72. PMID 16244520
- [Background] Wilson RD, Bennett ME, Lechman TE, Stager KW, Chae J. Single-lead percutaneous peripheral nerve stimulation for the treatment of hemiplegic shoulder pain: a case report. Arch Phys Med Rehabil. 2011 May;92(5):837-40. doi: 10.1016/j.apmr.2010.11.003. PMID 21530732
- [Background] Yu DT, Chae J, Walker ME, Fang ZP. Percutaneous intramuscular neuromuscular electric stimulation for the treatment of shoulder subluxation and pain in patients with chronic hemiplegia: a pilot study. Arch Phys Med Rehabil. 2001 Jan;82(1):20-5. doi: 10.1053/apmr.2001.18666. PMID 11239281
- [Background] Yu DT, Chae J, Walker ME, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Frost FS, Grill JH, Feldstein M, Fang ZP. Intramuscular neuromuscular electric stimulation for poststroke shoulder pain: a multicenter randomized clinical trial. Arch Phys Med Rehabil. 2004 May;85(5):695-704. doi: 10.1016/j.apmr.2003.07.015. PMID 15129391
- [Background] Yu DT, Chae J, Walker ME, Hart RL, Petroski GF. Comparing stimulation-induced pain during percutaneous (intramuscular) and transcutaneous neuromuscular electric stimulation for treating shoulder subluxation in hemiplegia. Arch Phys Med Rehabil. 2001 Jun;82(6):756-60. doi: 10.1053/apmr.2001.23310. PMID 11387579
- [Background] Koog YH, Jin SS, Yoon K, Min BI. Interventions for hemiplegic shoulder pain: systematic review of randomised controlled trials. Disabil Rehabil. 2010;32(4):282-91. doi: 10.3109/09638280903127685. PMID 20055567
- [Background] Snels IA, Beckerman H, Lankhorst GJ, Bouter LM. Treatment of hemiplegic shoulder pain in the Netherlands: results of a national survey. Clin Rehabil. 2000 Feb;14(1):20-7. doi: 10.1191/026921500668239146. PMID 10688341
- [Background] Soo Hoo J, Paul T, Chae J, Wilson RD. Central hypersensitivity in chronic hemiplegic shoulder pain. Am J Phys Med Rehabil. 2013 Jan;92(1):1-9; quiz 10-3. doi: 10.1097/PHM.0b013e31827df862. PMID 23255268
- [Background] Wilson RD, Harris MA, Gunzler DD, Bennett ME, Chae J. Percutaneous peripheral nerve stimulation for chronic pain in subacromial impingement syndrome: a case series. Neuromodulation. 2014 Dec;17(8):771-6; discussion 776. doi: 10.1111/ner.12152. Epub 2014 Feb 11. PMID 24512114
- [Background] Wilson RD, Harris MA, Bennett ME, Chae J. Single-lead percutaneous peripheral nerve stimulation for the treatment of shoulder pain from subacromial impingement syndrome. PM R. 2012 Aug;4(8):624-8. doi: 10.1016/j.pmrj.2012.03.002. PMID 22920317
- [Background] Paul TM, Soo Hoo J, Chae J, Wilson RD. Central hypersensitivity in patients with subacromial impingement syndrome. Arch Phys Med Rehabil. 2012 Dec;93(12):2206-9. doi: 10.1016/j.apmr.2012.06.026. Epub 2012 Jul 10. PMID 22789774
- See also: Cleveland FES Center — http://fescenter.org/index.php
- See also: The MetroHealth System - Clinical Trials — http://www.metrohealth.org

RESULTS

PARTICIPANT FLOW:
Groups:
- PNS + PT: The PNS+PT Group will receive peripheral nerve stimulation treatment for three weeks (6 hours daily) with an Intramuscular Electrical Stimulator following a 1 week electrode stabilization period,and also receive eight 60-minute sessions of outpatient physical therapy focused on shoulder pain over the same 4 week period. Peripheral Nerve Stimulation: The stimulation system includes an external stimulator, percutaneous lead and pad. The stimulator snaps onto the pad. The pad serves as the anode. The 1-channel stimulator outputs a biphasic current waveform with current pulse parameter ranges suitable for PNS. The percutaneous lead is inserted using an introducer (like a hypodermic needle) which is withdrawn and the lead is retained in the muscle by a barb at its tip. After a 1-week stabilization period, stimulation is initiated (6 hrs/day). The duty cycle and daily dose remain constant, but stimulus parameters may be adjusted by the research staff as deemed appropriate. The treatment period is 3 weeks after which the lead will be removed. Total time of electrode implantation is no more than 29 days. Physical Therapy: Participants will receive 8 60-minute sessions of outpatient therapy over a 4 week period concurrent with PNS or sham-PNS treatment. Therapy may include: Proper Positionand Handling, Therapeutic positioning and Strengthening Exercises, Mirror Therapy, Task-specific Therapy, Home Exercise Program, and a Mental Practice program.
- PNS + Sham-PT: The PNS + sham-PT Group will receive peripheral nerve stimulation treatment for 3weeks (6 hours daily) with an Intramuscular Electrical Stimulator following a 1week electrode stabilization period, and also receive eight 60-minute sessions of sham outpatient physical therapy not focused on shoulder pain over the same four week period. Peripheral Nerve Stimulation: The stimulation system includes an external stimulator, percutaneous lead and pad. The stimulator snaps onto the pad. The pad serves as the anode. The 1-channel stimulator outputs a biphasic current waveform with current pulse parameter ranges suitable for PNS. The percutaneous lead is inserted using an introducer (like a hypodermic needle) which is withdrawn and the lead is retained in the muscle by a barb at its tip. After a 1-week stimulation is initiated (6 hrs/day). The duty cycle and daily dose remain constant, but stimulus parameters may be adjusted by the research staff as appropriate. The treatment period is 3 weeks after which the lead is removed. Total time of electrode implantation is no more than 29 days. Sham-PT: Participants randomized to sham-PT will receive 8 60-minute sessions with therapists with the goal of controlling for the effect of regular contact with a therapist in a therapeutic environment. Therapists will provide sham ultrasound therapy and light application of inert gel to the shoulder for 10 minutes, Pre-Gait Training or Gait training, Exercise therapy, and relaxation therapy.
Period: Overall Study
Arm/Group | PNS + PT | PNS + Sham-PT | Sham-PNS + PT
Started | 31 | 32 | 33
Completed | 27 | 26 | 25
Not Completed | 4 | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- PNS + PT: The PNS+PT Group will receive peripheral nerve stimulation treatment for three weeks (6 hours daily) with an Intramuscular Electrical Stimulator following a 1 week electrode stabilization period,and also receive eight 60-minute sessions of outpatient physical therapy focused on shoulder pain over the same 4 week period. Peripheral Nerve Stimulation: The stimulation system includes an external stimulator, percutaneous lead and pad. The stimulator snaps onto the pad. The pad serves as the anode. The 1-channel stimulator outputs a biphasic current waveform with current pulse parameter ranges suitable for PNS. The percutaneous lead is inserted using an introducer (like a hypodermic needle) which is withdrawn and the lead is retained in the muscle by a barb at its tip. After a 1-week stabilization period, stimulation is initiated (6 hrs/day). The duty cycle and daily dose remain constant, but stimulus parameters may be adjusted by the research staff as deemed appropriate. The treatment period is 3 weeks after which the lead will be removed. Total time of electrode implantation is no more than 29 days. Physical Therapy: Participants will receive 8 60-minute sessions of outpatient therapy over a 4 week period concurrent with PNS or sham-PNS treatment. Therapy may include: Proper Position and Handling, Therapeutic positioning and Strengthening Exercises, Mirror Therapy, Task-specific Therapy, Home Exercise Program, and a Mental Practice program.
- Total: Total of all reporting groups
Arm/Group | PNS + PT | PNS + Sham-PT | Sham-PNS + PT | Total
Number analyzed (Participants) | 31 | 32 | 33 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 24 | 23 | 76
  >=65 years | 2 | 8 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (8.4) | 59.5 (9.6) | 58.9 (9.9) | 58.2 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 13 | 36
  Male | 21 | 19 | 20 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 11 | 15 | 43
  White | 13 | 20 | 14 | 47
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 33 | 96
Short Form (SF) Question 3 (BPI-SF3) absolute value [Mean (Full Range); unit: units on a scale] — The BPI has excellent psychometrics and is recommended for the assessment of pain in clinical trials. The developers of the BPI recommend BPI SF-3, the "pain worst" rating, as the primary response metric. The question asks participants to rate their worst pain in the prior 7-d on a 0 to 10 numeric rating scale, where "0" indicates "No pain" and "10" indicates "Pain as bad as you can imagine." Lower score means better outcome Absolute values are reported at Baseline. Worst Pain in the Last Week (0-10), 95% CI
  units on a scale | 7.129 [6.1 to 8.2] | 7.406 [6.4 to 8.4] | 8.061 [7.1 to 9.1] | 7.542 [6.1 to 9.1]

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (BPI)- Short Form (SF) Question 3 (BPI-SF3) - Mean Change From Baseline
Description: Brief Pain Inventory Short Form 3: The BPI has excellent psychometrics and is recommended for the assessment of pain in clinical trials. The developers of the BPI recommend BPI SF-3, the "pain worst" rating, as the primary response metric. The question asks participants to rate their worst pain in the prior 7-d on a 0 to 10 numeric rating scale, where "0" indicates "No pain" and "10" indicates "Pain as bad as you can imagine." Lower score means better outcome Baseline is absolute value and change value is reported for 4 weeks, 16 weeks and 28 weeks.
Time Frame: Baseline, 4 weeks(end of treatment), 16 weeks, 28 weeks
Population: Some participants drop out, withdraw consent, or are lost before later visits or assessments.
  Their later data points are missing, so they're not included in analyses for those timepoints.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PNS + PT | PNS + sham-PT | sham-PNS + PT
Number analyzed (Participants) | 31 | 32 | 33
units on a scale
  Baseline (absolute Value) | 7.1 [6.1 to 8.1] | 7.4 [6.4 to 8.4] | 8.1 [7.1 to 9.1]
  End of Treatment (change value): number analyzed (Participants) | 31 | 31 | 31
  End of Treatment (change value) | -2.8 [-3.9 to -1.8] | -2.4 [-3.4 to 1.4] | -2.4 [-3.4 to -1.4]
  16 weeks (change value): number analyzed (Participants) | 29 | 29 | 28
  16 weeks (change value) | -3.9 [-5.0 to -2.9] | -2.4 [-3.4 to -1.4] | -2.9 [-4.0 to -1.9]
  28 weeks (change value): number analyzed (Participants) | 28 | 27 | 26
  28 weeks (change value) | -2.8 [-4.3 to -1.4] | -2.1 [-3.2 to -1.0] | -3.1 [-4.0 to -2.0]

2. Other Pre Specified Outcome: Adverse Events (Number of Participants With Related Adverse Events)
Description: Related adverse events are documented as Safety data.
Time Frame: Week 2 - Week 5
Population: All subject who completed Baseline, Treatment and End of treatment assessments are included in the related adverse events reporting
Measure: Count of Participants; unit: Participants
Arm/Group | PNS + PT | PNS + sham-PT | sham-PNS + PT
Number analyzed (Participants) | 31 | 32 | 33
Participants | 13 | 15 | 14

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over the duration of the study of ~ 7 months
Arm/Group | PNS + PT | PNS + Sham-PT | Sham-PNS + PT
All-Cause Mortality (participants affected / at risk) | 1/31 | 0/32 | 1/33
Serious Adverse Events (participants affected / at risk) | 2/31 | 3/32 | 5/33
Other Adverse Events (participants affected / at risk) | 19/31 | 21/32 | 16/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PNS + PT (N=31) | PNS + Sham-PT (N=32) | Sham-PNS + PT (N=33)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Event (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Kidney Stones (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PNS + PT (N=31) | PNS + Sham-PT (N=32) | Sham-PNS + PT (N=33)
Retained Lead Fragment after Lead explant (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 4 (4)
Accidental Dislodgement of Lead (Surgical and medical procedures) | 2 (2) | 2 (2) | 4 (4)
Pain, related or possible related (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Skin Irritation, related or possible related (Skin and subcutaneous tissue disorders) | 13 (13) | 16 (16) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT02893267/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT02893267/SAP_001.pdf